CLINICAL TRIAL: NCT06163651
Title: Promoting Parent and Child Well-Being and Reducing the Need for Foster Care: An Evaluation of a One-Year, Home-Visiting and Case Management Program for People Using Substances
Brief Title: Evaluating a One-Year Version of the Parent-Child Assistance Program
Acronym: PCAP-1
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oklahoma (Other)
Collaborators: Children's Bureau - Administration for Children and Families (Other); Oklahoma Department of Health and Human Services (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 90FA3011
Record Dates: First submitted 2023-11-20; First posted 2023-12-11 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-06

CONDITIONS: Alcohol Use Disorder; Substance Use Disorders; Alcohol Use Complicating Pregnancy, Unspecified Trimester; Drug Use Disorders; Drug Use Complicating Pregnancy, Unspecified Trimester
Keywords: Parent-Child Assistance; Substance Use Disorder; Addictions; Drug Dependence; Drug Abuse; Alcohol Dependence; Alcohol Abuse; Alcoholism; Recovery Services; PCAP
MeSH Terms: conditions — Alcoholism; Substance-Related Disorders; Behavior, Addictive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment Group (Experimental): The treatment group consists of parents who meet our eligibility criteria. Parents in the treatment group will receive PCAP-1 services through the work of highly trained, closely-supervised case managers.
  Interventions: Behavioral: Parent-Child Assistance Program - One-Year Version
- Control Group (No Intervention): The control group consists of parents who meet our eligibility criteria and are part of administrative data from the Oklahoma Department of Human Services in a comparable county to our intervention county, or from prior historical cases within the same county. Parents in the control group can access "services as usual" in the community, but will not receive PCAP in any form.

INTERVENTIONS:
Behavioral: Parent-Child Assistance Program - One-Year Version — Case managers work closely with parents over the course of one year, meeting them in their own homes when possible, to help them set goals and take advantage of available resources.
  Arms: Treatment Group

SUMMARY:
The proposed project seeks to achieve three objectives that will, collectively, evaluate the effectiveness of a one-year version of the Parent-Child Assistance Program (PCAP-1) -a model for a home visitation and case management program for parents who used substances. First, the proposed project aims to estimate the causal impact of PCAP-1 on preventing the need for foster care and promoting reunification. Second, the project will estimate PCAP-1's effectiveness in achieving other program goals: parent recovery, parent's connection with needed comprehensive community resources, and preventing future children from being exposed to drugs and alcohol. Finally, causal evidence of program effectiveness across the prior two objectives would enable PCAP-1 to be rated according to strength of evidence on relevant federal registries (i.e., FFPSA and HOMEVEE). All objectives will be pursued with substantial backing from public and private partners, including the Oklahoma Department of Human Services (OK's Title IV-E agency). This quasi-experimental project will recruit 40 new participants to receive one year of PCAP-1 services. It will use administrative data on participants from the Oklahoma Department of Human Services for the control group. Given that the population PCAP serves are disproportionately poor and low-income and PCAP is designed to be culturally competent and relevant, PCAP-1 harbors the potential to address inequities in child welfare outcomes, substance use disorder treatment services, and child and family well- being by improving outcomes for these families. With a strong backing by state agencies and community partners, the evaluation of PCAP-1 will contribute to a knowledge gap in the field for in-home program models serving a highly vulnerable population with high rates of child welfare involvement and use of foster care.

DETAILED DESCRIPTION:
PCAP is a three-year, intensive case management intervention for pregnant and postpartum individuals who have used substances during their current or most recent pregnancy. PCAP provides mothers with a case manager with whom they meet biweekly, in the home or in other community settings. Case managers coach mothers in setting their own goals and taking steps to achieve them, provide practical assistance, serve as role models, and offer emotional support and encouragement. They connect mothers to community resources and recovery supports tailored to the participant's needs and goals. On average, case managers carry a caseload of 16 mothers/families, receive at least biweekly individual clinical supervision by a master's-level clinician, biweekly group supervision, and individual consultation with their supervisor whenever needed. Case managers work with the mother and the child with prenatal substance exposure and other family members in support of the participant's goals and recovery.

This project seeks to evaluate a one-year version of PCAP (PCAP-1), aligned with the time frame of the FFPSA federal matching funds for prevention programs with evidence of effectiveness. PCAP was originally designed to be a three-year intervention as it was theorized that three years comprised a realistic time frame during which a mother can form a strong therapeutic alliance with a case manager and undergo the developmental process of making gradual behavioral changes. Indeed, for many clients, who may never have known the steady presence of a trusted parent or other individual in their lives, the beginning of that process is slow and tentative. The three-year duration was also chosen to provide clients with ample time to make fundamental changes in their lives. In the standard PCAP program, preparing for post-intervention does not begin until Year 3. The investigators now theorize that the most significant changes happen within the first year, and a one-year program may be a better fit for many clients, especially those who are child welfare-involved. A shorter duration may also serve as an external motivator to clients in completing their goals, as they will know they have a one-year time frame during which they will have assistance, and they will sooner begin anticipating the post-intervention period. A one-year intervention is also indicated under the parameters of the FFPSA as the FFPSA provides matching funds for one year of evidence-based in-home services to child welfare-involved families to prevent the need for foster care.

The specific objectives of this project are to:

1. Establish causal evidence of effectiveness of PCAP-1 in preventing the need for foster care and promoting reunification
2. Establish causal evidence of the effectiveness of PCAP-1 in achieving other key goals: (a) Parent achieves and stays in recovery, (b) Parent accesses comprehensive services to meet needs to achieve and maintain a healthy family life
3. Lay the groundwork to be rated by relevant federal registries according to strength of the program's evidence of effectiveness for purposes of sustainability, spread, and replication.

In 2021, PCAP and a rigorous randomized controlled trial (RCT) testing the benefits of the program was implemented in Oklahoma. Two Oklahoma sites began enrolling clients in late 2022. Each site will enroll 100 participants, randomly assigned to the experimental groups: treatment and control (services as usual). The project proposed herein will complement the ongoing RCT but offers the important additional benefit of adapting and extending PCAP to a third study site and evaluating a one-year version of PCAP. This adaptation is important because client and case manager mindsets and priorities may be very different when faced with a one-year time frame rather than a three-year time frame. Furthermore, a one-year version of PCAP is more consistent with the Adoption and Safe Families Act timelines for permanency hearings to start to establish the permanency plan for a child in foster care.

Using the recruitment strategies described above, 40 eligible people will be recruited into PCAP-1 from an additional PCAP site. The one-year intervention will take place over the three-year project period, with enrollment into PCAP-1 occurring on a rolling basis over the first two years of this study. Two case managers will each be assigned 20 PCAP-1 participants over the study period to avoid the n=1 confounding problem.

This quasi-experimental design incorporates a control group to compare one-year outcomes with the PCAP-1 participants. The approximately 40 people making up the control group will come from the administrative data provided by the Oklahoma Department of Human Services. The control group will be matched with the PCAP-1 treatment group based on characteristics such as age, race/ethnicity, and socioeconomic status.

The Self-Administered Survey (SAS) will capture outcome data about individuals in PCAP-1. The SAS was developed by the investigator team drawing primarily upon standardized scales and measures used in addictions research and related subfields that have solid psychometric properties. Many of these standardized scales and measures have also been found to be valid measures for use in diverse populations. The investigators took these studies into account when selecting our measures. Information from the SAS is secondary to our 3 main research objectives and questions. However, the research team is proposing to collect this information for the PCAP-1 evaluation as it broadens the outcomes examined, maximizes the research investment, and allows us to also report on important other outcomes in addictions research, as well as examine mechanisms of success. The SAS elicits information from clients along several dimensions covering a wide range of client behavior metrics and social psychological concepts important for addiction research, including criminal justice involvement, additional adverse childhood experiences (ACEs) from an expanded ACEs instrument, social support, mental health, self- efficacy, addiction beliefs, parenting practices, and parent/child experiences. These measures allow us to examine both predictors of success, as well as additional outcomes stemming from the intervention. The SAS will be administered to all study participants at baseline and at 12 and 18 months following baseline.

Additionally, PCAP case managers will complete a standardized questionnaire regarding each of their clients (treated participants) at 6 and 12 months. These biannual case-manager reports characterize clients' substance use and SUD treatment; child custody and child welfare involvement; family planning and pregnancy; connection to services for client, child/ren, and other family members; housing; income and employment; education; and criminal justice involvement. Shorter monthly reports will document whether the client and index child were seen and, if not, efforts to reach the client; substance use and SUD treatment; and child custody and child welfare involvement.

Moreover, this project's state agency partnership will also contribute complementary child welfare administrative data to the evaluation of PCAP-1. OK DHS maintains the Statewide Automated Child Welfare Information System, commonly referred to as KIDS. The KIDS data system contains an entry for each referral or action incident regarding potential child neglect or abuse. These referral records contain a wealth of information about the referred child, the primary and secondary caregivers, and the nature and outcome of the referral. Regarding the referred child, the records contain information on demographics, measures of mental and physical health, an assessment of child safety, and education. For caregivers, the KIDS system contains information on demographics, criminal justice system involvement, employment and income, and receipt of public assistance, among other data elements. In terms of the nature and outcome of the referral, KIDS contains information on the reason for the referral as well as its disposition. The data contain detailed information on removals, placement into foster care, and subsequent placements over time. Finally, the records indicate whether and when the child was reunified with the original caregiver after removal. These data will allow us to document child removals and reunifications, in the context of child safety (from recurrence of maltreatment).

ELIGIBILITY:
Inclusion Criteria:

* People over the age of 18
* Parents with children under the age of 6 living with them
* Resides within a 50-mile radius of Enid, OK or Oklahoma City, OK (for treatment group)

Exclusion Criteria:

- Incarcerated at the time of enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-06-23 (Actual); Primary Completion 2026-09-29 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Proportion of target children not placed in foster care | Measured after 1 year of study participation.
  The target child is not placed in foster care.
Parent acquires or maintains child custody | Measured after 1 year of study participation.
  The parent has physical custody of the target child.
Reduction in costs to state agencies | Measured after 1 year of study participation.
  Reduced costs to state agencies following PCAP-1 participation.

SECONDARY OUTCOMES:
Proportion of parents who acquire or maintain stable housing | Measured after 1 year of study participation.
  The parent resides in stable housing.
Proportion of parents who acquire or maintain employment | Measured after 1 year of study participation.
  The parent is employed.
Proportion of parents who enroll in or complete an educational program | Measured after 1 year of study participation.
  The parent has completed or is enrolled in an educational program.
Proportion of parents who receive public benefits | Measured after 1 year of study participation.
  The parent receives public benefits (e.g., housing, food, cash)
Proportion of parents with ongoing criminal justice involvement | Measured after 1 year of study participation.
  The parent has had new involvement with the criminal justice system.

CONTACTS AND LOCATIONS:
Overall Officials: Julie Gerlinger, PhD, Principal Investigator — University of Oklahoma; Erin Maher, PhD, Principal Investigator — University of Oklahoma; Susan Stoner, PhD, Principal Investigator — University of Washington
Locations (2):
- United States (2):
  - Remote Worker, Enid, Oklahoma
  - Remote Worker, Oklahoma City, Oklahoma

IPD SHARING:
Plan to Share IPD: No